CLINICAL TRIAL: NCT06230640
Title: Evaluation of TEG 6S Platelet Mapping® During Cardiopulmonary Bypass for Cardiac Surgery to Detect Postoperative Biological Coagulopathy
Brief Title: Evaluation of TEG 6S PM® During Cardiopulmonary Bypass to Detect Postoperative Biological Coagulopathy
Acronym: PREDIPOC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0167
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Coagulopathy; Cardiopulmonary Bypass; Cardiac Surgery
Keywords: Coagulopathy; cardiac surgery; cardiopulmonary bypass
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac surgery with cardiopulmonary bypass: Any subject undergoing cardiac surgery with cardiopulmonary bypass and at high risk of bleeding and transfusion.
  Interventions: Diagnostic Test: In vitro medical diagnostic device TEG6s® Platelet Mapping

INTERVENTIONS:
Diagnostic Test: In vitro medical diagnostic device TEG6s® Platelet Mapping — Preoperative period:
  * Pre-operative blood sampling, according to the usual practices of the unit before surgery
  * Collection of the patient's usual demographic characteristics
  per operative period :
  * After anesthetic induction:a TEG6S platelet mapping® sampled from the arterial catheter routinely placed after anesthetic induction
  * During the CPB, 30 min before aortic declamping: performing TEG 6S platelet mapping® (heparinized tube)
  * 5 min after heparin antagonization by protamine, after the weaning of the bypass, and before any transfusion: performing a TEG 6S citrate® (citrated tube)
  Post-operative period (resuscitation):
  • postoperative bleeding at 2 hours and during the first 12 hours.
  Other Names: Comparison between TEG 6S platelet mapping® and TEG 6S global hemostasis Assessment of platelet inhibition rate

SUMMARY:
This is a prospective study to evaluate the predictive value of the TEG 6s platelet mapping® (TEG 6s® PM) performed during cardiopulmonary bypass (CPB) in the prediction of biological coagulopathy (determined by TEG 6S global hemostasis®), in cardiac surgery with high risk of bleeding.

DETAILED DESCRIPTION:
The aim of this prospective study is to evaluate the predictive value of the R time (HKH) given by the TEG 6s platelet mapping® performed during the CPB in the prediction of postoperative biological coagulopathy.

In order to evaluate its interest and to validate its use during cardiac surgery with high bleeding risk under CPB, we plan to compare 2 thromboelastographic tests in the detection of biological coagulopathy: TEG 6S citrated® (reference) and TEG 6S platelet mapping®. Biological coagulopathy is defined by a kaolin-heparinase assay coagulation/reaction time (CKH R) value of 7 min on TEG 6S citrated® (fibrinogen impairment defined by a Comparison of functional fibrinogen Maximal Amplitude (CFF MA) < 20 mm, and CKH MA impairment (< 60 mm), in accordance with established laboratory standard values.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Cardiac surgery under cardiopulmonary bypass with high risk of bleeding defined among:
* CPB with circulatory arrest
* cardiac transplantation
* Redo surgery
* infective endocarditis
* predicted duration of CBP ≥ 120 min
* High transfusion risk defined by a Trust predictive score ≥ 3 (Transfusion Risk Understanding Scoring Tool)

Exclusion Criteria:

* Patient with heparin allergy or heparin-induced thrombocytopenia
* Use of direct oral anticoagulant (DAA) with anti-factor X activity (Apixaban, Rivaroxaban) < 72h, even if antagonized
* Patient on partially or fully antagonized VKAs
* Opposition to participation after a period of reflection
* Adult protected by law (guardianship, curatorship)
* Person deprived of liberty
* Person participating in another study with an exclusion period still in progress
* Patient not affiliated to a social security scheme or not benefiting from such a scheme
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject undergoing cardiac surgery with cardiopulmonary bypass circulation and at high risk of bleeding and transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Prolongation of the R in kaolin with heparinase (HKH) of TEG 6S platelet mapping® during cardiopulmonary bypass. | After anesthetic induction; 30 min before aortic declamping and 5min after antagonization
  The measurement of the R time (coagulation time in minutes) is automated by using a TEG 6S® analyzer from the Haemonetics laboratory and using the TEG 6S platelet mapping® and global hemostasis® cartridge.

SECONDARY OUTCOMES:
Change in maximum amplitude HKH (MA HKH) of TEG 6S platelet mapping® during CPB. | After anesthetic induction; 30 min before aortic declamping
  The measurement of the various parameters (coagulation time R in minutes, maximum amplitude of the clot strength MA in millimeter mm) is automated by using a TEG 6S® analyzer from the Haemonetics laboratory, which is already available in our unit, and using the TEG 6S platelet mapping® and citrated® cartridge.
Change in maximum amplitude in the presence of fibrinogen activator (MA ActF) of TEG 6S platelet mapping® during CPB. | After anesthetic induction; 30 min before aortic declamping
  The measurement of the various parameters (coagulation time R in minutes, maximum amplitude of the clot strength MA in millimeter mm) is automated by using a TEG 6S® analyzer from the Haemonetics laboratory, which is already available in our unit, and using the TEG 6S platelet mapping® and citrated® cartridge.
Maximum amplitude change in the presence of arachidonic acid (MA AA) in TEG 6S platelet mapping® during CPB. | After anesthetic induction; 30 min before aortic declamping
  The measurement of the various parameters (coagulation time R in minutes, maximum amplitude of the clot strength MA in millimeter mm) is automated by using a TEG 6S® analyzer from the Haemonetics laboratory, which is already available in our unit, and using the TEG 6S platelet mapping® and citrated® cartridge.
Maximum amplitude change in the presence of P2Y12 receptor activating ADP (MA ADP) of TEG 6S platelet mapping® during CPB. | After anesthetic induction; 30 min before aortic declamping
  The measurement of the various parameters (coagulation time R in minutes, maximum amplitude of the clot strength MA in millimeter mm) is automated by using a TEG 6S® analyzer from the Haemonetics laboratory, which is already available in our unit, and using the TEG 6S platelet mapping® and citrated® cartridge.
Correlation between the R HKH time of TEG 6S platelet mapping® and the R CKH of TEG 6S citrated®. | After anesthetic induction; 30 min before aortic declamping and 5min after antagonization
  The measurement of the various parameters (coagulation time R in minutes, maximum amplitude of the clot strength MA in millimeter mm) is automated by using a TEG 6S® analyzer from the Haemonetics laboratory, which is already available in our unit, and using the TEG 6S platelet mapping® and citrated® cartridge.
Post-operative bleeding over the first 2 hours | during the 2 hours post-surgery
  Volume measured by drains connected to graduated sterile jars. Blood volume in milliliters (mL)
Post-operative bleeding over 12 hours in intensive care | during the 12 hours post-surgery
  Volume measured by drains connected to graduated sterile jars. Blood volume in milliliters (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bourdois, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Département d'Anesthésie Réanimation cardio-thoracique - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yamamoto Y, Sato Y, Takahashi M, Yamamoto H, Echizen M, Uchida T. TEG6s Platelet Mapping assay for the estimation of plasma fibrinogen concentration during cardiovascular surgery: a single-center prospective observational study. J Anesth. 2022 Feb;36(1):79-88. doi: 10.1007/s00540-021-03009-4. Epub 2021 Oct 13. PMID 34643817